CLINICAL TRIAL: NCT06002048
Title: AI Ready and Exploratory Atlas for Diabetes Insights
Acronym: AI-READI
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Aaron Y Lee, Associate Professor, Department of Ophthalmology, University of Washington
Other Study IDs: STUDY00016228; 3OT2OD032644-01S3 (NIH)
Record Dates: First submitted 2023-07-24; First posted 2023-08-21 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes
Keywords: Machine Learning; Type 2 Diabetes; Retinal Imaging; Data Sharing; Equitable Data Collection
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Healthy: Participants who do not have Type 1 or Type 2 Diabetes
- Pre-diabetes/Diet Controlled: Participants with pre-Type 2 Diabetes and those with Type 2 Diabetes whose blood sugar is controlled by diet
- Oral Medication and/or Non-insulin-injectable Medication Controlled: Participants with Type 2 Diabetes whose blood sugar is controlled by oral or injectable medications other than insulin
- Insulin Dependent: Participants with Type 2 Diabetes whose blood sugar is controlled by insulin

SUMMARY:
The study will collect a cross-sectional dataset of 4000 people across the US from diverse racial/ethnic groups who are either 1) healthy, or 2) belong in one of the three stages of diabetes severity (pre-diabetes/diet controlled, oral medication and/or non-insulin-injectable medication controlled, or insulin dependent), forming a total of four groups of patients. Clinical data (social determinants of health surveys, continuous glucose monitoring data, biomarkers, genetic data, retinal imaging, cognitive testing, etc.) will be collected. The purpose of this project is data generation to allow future creation of artificial intelligence/machine learning (AI/ML) algorithms aimed at defining disease trajectories and underlying genetic links in different racial/ethnic cohorts. A smaller subgroup of participants will be invited to come for a follow-up visit in year 4 of the project (longitudinal arm of the study). Data will be placed in an open-source repository and samples will be sent to the study sample repository and used for future research.

DETAILED DESCRIPTION:
The Artificial Intelligence Ready and Exploratory Atlas for Diabetes Insights (AI-READI) project seeks to create a flagship ethically-sourced dataset to enable future generations of artificial intelligence/machine learning (AI/ML) research to provide critical insights into type 2 diabetes mellitus (T2DM), including salutogenic pathways to return to health. The ability to understand and affect the course of complex, multi-organ diseases such as T2DM has been limited by a lack of well-designed, high quality, large, and inclusive multimodal datasets. The AI-READI team of investigators will aim to collect a cross-sectional dataset of 4,000 people and longitudinal data from 10% of the study cohort across the US. The study cohort will be balanced for self-reported race/ethnicity, gender, and diabetes disease stage. Data collection will be specifically designed to permit downstream pseudo-time manifold analysis, an approach used to predict disease trajectories by collecting and learning from complex, multimodal data from participants with differing disease severity (normal to insulin-dependent T2DM). The long-term objective for this project is to develop a foundational dataset in T2DM, agnostic to existing classification criteria or biases, which can be used to reconstruct a temporal atlas of T2DM development and reversal towards health (i.e., salutogenesis). Six cross-disciplinary project modules involving teams located across eight institutions will work together to develop this flagship dataset. Data will be optimized for downstream AI/ML research and made publicly available. This project will also create a roadmap for ethical and equitable research that focuses on the diversity of the research participants and the workforce involved at all stages of the research process (study design and data collection, curation, analysis, and sharing and collaboration).

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 40 years old)
* Patients with and without type 2 diabetes
* Able to provide consent
* Must be able to read and speak English

Exclusion Criteria:

* Adults older than 85 years of age
* Pregnancy
* Gestational diabetes
* Type 1 diabetes

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients will be recruited into one of four groups: 1) healthy/no diabetes, 2) pre-diabetes/borderline diabetes/diet-controlled diabetes, 3) oral medication and/or non-insulin injectable medication controlled type 2 diabetes, or 4) insulin dependent type 2 diabetes. The investigators aim to recruit approximately 1000 patients into each of the four groups. Patients will be recruited from University of Washington (UW), University of California at San Diego (UCSD), and University of Alabama at Birmingham (UAB). The study aims to recruit 1,000 subjects from each of the following racial and ethnic groups: white, Asian, Hispanic, and Black. Subjects will be age- and sex-matched within and between groups.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Best-corrected visual acuity | July 19, 2023-January 1, 2027
  Both photopic and mesopic for right and left eyes individually
Contrast Sensitivity | July 19, 2023-January 1, 2027
  Both photopic and mesopic for right and left eyes individually
Optical coherence tomography (OCT) | July 19, 2023-January 1, 2027
fundus photography | July 19, 2023-January 1, 2027
fluorescence lifetime imaging ophthalmoscopy (FLIO) | July 19, 2023-January 1, 2027
optical coherence tomography angiography (OCTA) | July 19, 2023-January 1, 2027
Continuous Glucose Monitoring | July 19, 2023-January 1, 2027
  Participants wear the Dexcom G6 Pro for 10 days
Home humidity | July 19, 2023-January 1, 2027
Home temperature | July 19, 2023-January 1, 2027
  measured in Fahrenheit
Volatile Organic Compounds (VOC) in home | July 19, 2023-January 1, 2027
Fine particulate matter that are 2.5 microns or less in diameter (PM2. 5) in home | July 19, 2023-January 1, 2027
Montreal Cognitive Assessment (MoCA) | July 19, 2023-January 1, 2027
  Testing memory and cognitive function. Scores range from 0-30, with scores above 26 indicating normal functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Lee, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - UC San Diego, San Diego, California
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No